CLINICAL TRIAL: NCT01933958
Title: Drug Use Investigation of Regorafenib/ STIVARGA for Gastrointestinal Stromal Tumor Progressed After Cancer Chemotherapy
Brief Title: Regorafenib Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16732; STIVARGA-GIST-01 (Other: company internal)
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Regorafenib; Gastrointestinal stromal tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with Regorafenib under practical manner for gastrointestinal stromal tumors progressed after cancer chemotherapy.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — The usual dosage is 160 mg of Regorafenib/ STIVARGA taken orally after meal once daily for 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks.

SUMMARY:
The objective of this study is to assess safety and effectiveness of Regorafenib using in real clinical practice

DETAILED DESCRIPTION:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Regorafenib for gastrointestinal stromal tumors progressed after cancer chemotherapy.

A total of 135 patients are to be enrolled and assessed in 6 months standard observational period. At 12 months and 24 months after the first administration of Regorafenib for confirmation of efficacy information including treatment duration and survival status of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Regorafenib/ STIVARGA and meet the product label.

Exclusion Criteria:

* Patients who are treated with Regorafenib/ STIVARGA and don't meet the product label.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are treated with Regorafenib/STIVARGA and meet the product label
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-09-04 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse drug reactions (ADRs) from the first administration of regorafenib. | Up to 6 months
Number of patients with serious adverse events(SAEs) from the first administration of regorafenib. | Up to 6 months
Number of Patients with serious adverse drug reactions (SADRs) from the first administration of Regorafenib | up to 6 months

SECONDARY OUTCOMES:
overall survival (OS) | Up to 3 years
time to treatment failure (TTF) | Up to 3 years
  TTF is defined as the time interval from start of Regorafenib/ STIVARGA therapy to the date of permanent discontinuation for any reason including disease progression, adverse event, patient preference or death.
tumour response | Up to 3 years
Integration analysis for safety in drug use investigations (DUIs) for both colorectal cancer and gastrointestinal stromal tumor. | Up to 3 years
  Integration analysis including incidence and risk factor of adverse drug reaction (ADR), serious adverse event (SAE) and serious adverse drug reaction (SADR)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, time point and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Komatsu Y, Muro K, Chosa M, Hirano K, Sunaya T, Ayukawa K, Hattori K, Nishida T. Large-scale, prospective observational study of regorafenib in Japanese patients with advanced gastrointestinal stromal tumors in a real-world clinical setting. Front Oncol. 2024 Jun 17;14:1412144. doi: 10.3389/fonc.2024.1412144. eCollection 2024. PMID 38952554
- [Derived] Komatsu Y, Doi T, Sawaki A, Kanda T, Yamada Y, Kuss I, Demetri GD, Nishida T. Regorafenib for advanced gastrointestinal stromal tumors following imatinib and sunitinib treatment: a subgroup analysis evaluating Japanese patients in the phase III GRID trial. Int J Clin Oncol. 2015 Oct;20(5):905-12. doi: 10.1007/s10147-015-0790-y. Epub 2015 Feb 6. PMID 25655899